CLINICAL TRIAL: NCT05366270
Title: Peripheral Neuroimmune Mechanisms of Hyperthermia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Simmie L. Foster, MD, Psychiatrist, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2019P001103; 5K23GM129630-03 (NIH)
Record Dates: First submitted 2022-04-18; First posted 2022-05-09 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Hyperthermia; Major Depressive Disorder; Inflammation
Keywords: Depression; Major Depressive Disorder; Inflammation; Hyperthermia; Mood Disorders
MeSH Terms: conditions — Hyperthermia; Depressive Disorder, Major; Inflammation; Depression; Mood Disorders

STUDY DESIGN:
Intervention Model Description: Subjects are randomized to Control/Sham and Intervention groups
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participant and clinician assessors will be blinded until study completion. The PI will only be unblinded in the event of an adverse event.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Whole Body Hyperthermia (WBH) (Experimental): A single treatment of Whole Body Hyperthermia will be administered using the Heckel Hyperthermia device. During this procedure, participants' core body temperature will be elevated to 38.5 degrees Celsius.
  Interventions: Device: WBH
- Sham (Sham Comparator): Under the sham condition, participants will enter the Heckel Hyperthermia device as in the active treatment condition, but will not receive the whole body hyperthermia treatment, and will instead only receive mild heating.
  Interventions: Device: Sham

INTERVENTIONS:
Device: WBH — Hyperthermia exposure using Heckel Hyperthermia Device
  Other Names: Whole Body Hyperthermia
  Arms: Whole Body Hyperthermia (WBH)
Device: Sham — Sham (mild heating) using Heckel Hyperthermia Device
  Arms: Sham

SUMMARY:
The goal of this study is to examine how whole-body hyperthermia affects the thermoinflammatory profile, which includes the combined immune and heat shock response, in patients with depression and whether these changes correlate with decreased depression in individuals with Major Depressive Disorder.

DETAILED DESCRIPTION:
The study is a maximum of 42-day randomized controlled trial (RCT) of Whole Body Hyperthermia (WBH) vs. Sham for subjects with depressive symptoms at the Depression Clinical Research Program (DCRP) at Massachusetts General Hospital (MGH). 60 subjects with Major Depressive Disorder (MDD), males and females, between the ages of 18 and 65 years will be recruited and undergo a screening visit prior to being randomized to receive a single treatment of WBH or sham. The primary endpoint will be measurement of Interleukin-6 (IL-6) and other inflammation associated proteins (cytokines and heat shock proteins) in the plasma at one hour, 24h and one-week post WBH. A further endpoint is treatment response defined by a decrease of 50% or more in the Inventory of Depressive Symptomatology, Clinician-Rated (IDS-CR) score at 7 days post-intervention, 2 weeks post-intervention, and 4 weeks post-intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Females and Males ages 18-65
2. English language proficiency
3. Ability to provide informed consent
4. Have a current primary psychiatric diagnosis of major depressive disorder (MDD) of at least 4 weeks duration, as defined by Diagnostic & Statistical Manual, 5th Edition (DSM-5) criteria using the MINI.
5. Score of ≥ 24 on the Inventory of Depressive Symptomatology - Clinician Rated (IDS-CR)
6. Individuals of childbearing potential must use an acceptable form of birth control.

Exclusion Criteria:

1. Pregnancy or planned pregnancy during study
2. Current breastfeeding
3. History of psychiatric hospitalization within the past year
4. Active suicidal intent ("yes" on item 4 or 5 on the Columbia-Suicide Severity Rating Scale)
5. History of bipolar disorder, psychotic disorders, eating disorders, and/or substance abuse or dependence (within the last year), as per the Mini-International Neuropsychiatric Interview (MINI)
6. Meeting DSM-5 criteria at screening for current obsessive compulsive disorder
7. A ≥25% drop in IDS-CR score from screen (V1) to baseline (V1b)
8. Positive urine toxicology screen due to illicit drug use or other exclusionary medications. (Potential false positives will be addressed on a case-by-case basis at the discretion of the investigator)
9. Serious unstable medical condition including cardiovascular, neurological, neoplastic, autoimmune, infectious or endocrine.
10. Morbid obesity (BMI > 40) and/or body shape that might increase the risk of cutaneous burning from the Heckel hyperthermia device (because of truncal skin being too close to the infrared lights).
11. Any history of or current diagnosis of thrombosis or thrombophilia; if it is unclear whether a subject has received this diagnosis, a signed release will be obtained to contact the subject's treating physician and obtain accurate diagnostic information. Depending on the recommendation of the treating physician, the subject may undergo appropriate testing with the treating physician to verify the diagnosis, and if the tests produce negative findings, the subject may be allowed to enter the study
12. Has a history of or an increased risk for gastrointestinal perforation such as a history of diverticulitis, stomach or intestinal ulcers or abdominal pain that does not go away
13. Using medication that might impact thermoregulatory capacity within 3 days of receiving WBH treatment, including: diuretics, barbiturates, beta-blockers, antipsychotic agents, anti-cholinergic agents or chronic use of antihistamines, aspirin (other than low-dose for prophylactic purposes), non-steroidal anti-inflammatory drugs (NSAIDs), systemic corticosteroids, or cytokine antagonists.
14. Use of any medication that could interact in such a way as to potentiate the sedative effect of lorazepam or ondansetron, or otherwise deemed unsafe per physician judgment.
15. Fever (Temp > 99) of unknown origin at the time of screen
16. Breast Implants
17. Unsafe cardiac status as defined by abnormal ECG reading at screening visit as determined by medical monitor, study doctor, or subject's primary care physician or cardiologist
18. Claustrophobia of sufficient severity to interfere with ability to enter/remain in Heckel device
19. A subject who in the opinion of the Principal Investigator would not be able to safely complete the study or would jeopardize study integrity

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Changes in serum levels of Interleukin-6 from baseline to post-treatment | baseline (pre-intervention), one hour post-intervention, 24 hours post-intervention, one week post-intervention
  Changes in serum levels of Interleukin-6 from baseline to post-treatment, measured by immunoassay
Decreases in depressive severity, as measured by the Inventory of Depressive Symptomatology, Clinician-Rated (IDS-CR) | baseline (pre-intervention), one week post-intervention, two weeks post-intervention, four weeks post-intervention
  The Inventory of Depressive Symptomatology is a valid and reliable 30-item measure that is designed to assess severity of depression. The questions focus on neurovegetative and other depressive symptoms experienced over the past seven days. Possible values range from 0 to 84, with lower scores indicating lower depressive severity. A decrease of 50% or more in the IDS-CR score is considered to be a positive response to treatment, while a final score of 11 or less is considered typical remission.
  Depressive severity will be measured at baseline and at three timepoints post-intervention using the IDS-CR.
Decreases in depressive severity, as measured by the Symptoms of Depression Questionnaire (SDQ) | baseline (pre-intervention), 24 hours post-intervention, one week post-intervention, two weeks post-intervention, four weeks post-intervention
  The Symptoms of Depression Questionnaire (SDQ) assesses irritability, anger attacks, and anxiety symptoms together with the commonly considered symptoms of depression. Depressive severity will be measured at baseline and at four timepoints post-intervention using the SDQ. Possible values range from 44 to 264, with lower scores indicating lower depressive severity.

SECONDARY OUTCOMES:
Changes in mental and physical functioning, as measured by the Patient Rated Outcome Measure Information System, 29-Item (PROMIS-29) | baseline (pre-intervention), one week post-intervention, two weeks post-intervention, four weeks post-intervention
  The PROMIS-29 is a short form assessment containing four items from each of seven domains (Depression, Anxiety, Physical Function, Pain Interference, Fatigue, Sleep Disturbance, and Ability to Participate in Social Roles and Activities) plus one pain intensity question (0-10 numeric rating scale). Possible values range from 4 to 20, with lower scores indicating better functioning.
Changes in mood, as measured by the Positive and Negative Affect Schedule (PANAS) | baseline (pre-intervention), 24 hours post-intervention, one week post-intervention, two weeks post-intervention, four weeks post-intervention
  The Positive and Negative Affect Schedule (PANAS) is a self-report measure that is made up of two mood scales, one measuring positive affect and the other measuring negative affect. Number of items: 10-items measuring positive affect, 10-items measuring negative affect. Scoring is broken down into a positive affect score and a negative affect score; possible values range from 10 to 50, with higher positive scores indicating higher positive affect, and higher negative scores indicating higher negative affect.
Changes to quality of life, as measured by the World Health Organization Wellbeing Index (WHO-5) | baseline (pre-intervention), one week post-intervention, two weeks post-intervention, four weeks post-intervention
  The World Health Organization-Five Well-Being Index (WHO-5) is a short self-reported measure of current mental wellbeing. Possible values range from 0 to 25, with lower scores indicating lower quality of life.
Changes to quality of life, as measured by the Quality of Life, Enjoyment, and Satisfaction Questionnaire | baseline (pre-intervention), one week post-intervention, two weeks post-intervention, four weeks post-intervention
  The Quality of Life Enjoyment and Satisfaction Questionnaire is a self-report measure designed to enable investigators to easily obtain sensitive measures of the degree of enjoyment and satisfaction experienced by subjects in various areas of daily functioning. Possible values range from 14 to 70, with lower scores indicating lower quality of life.
Reduction in perceived stress, as measured by the Perceived Stress Scale (PSS) | baseline (pre-intervention), one week post-intervention, two weeks post-intervention, four weeks post-intervention
  The Perceived Stress Scale (PSS) is the most widely used psychological instrument for measuring the perception of stress. It is a measure of the degree to which situations in one's life are appraised as stressful. Items were designed to tap how unpredictable, uncontrollable, and overloaded respondents find their lives. Possible values range from 0 to 40, with lower scores indicating lower levels of perceived stress.
Decreases in depressive severity, as measured by the Hamilton Depression Rating Scale 6-Item Self-Report (HAMD-6) | baseline (pre-intervention), 24 hours post-intervention, one week post-intervention, two weeks post-intervention, four weeks post-intervention
  The Hamilton Depression Rating scale (self-report, 6-item) is specific to the core depressive symptoms of depressed mood, guilt, work and activities, psychomotor retardation, psychic anxiety, and general somatic symptoms (energy and physical pain), and it is unidimensional. Possible values range from 0 to 22, with lower scores indicating lower levels of depressive severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital Depression Clinical & Research Program, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No